CLINICAL TRIAL: NCT06192446
Title: Factors Influencing Adherence to Adjuvant Endocrine Therapy in Women With Early Breast Cancer in Croatia
Brief Title: Factors Influencing Adherence to Adjuvant Endocrine Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zagreb (Other)
Responsible Party: Principal Investigator, Iva Mucalo, Associate professor at the Center for Applied Pharmacy., University of Zagreb
Other Study IDs: 380-130/134-22-4
Record Dates: First submitted 2023-12-07; First posted 2024-01-05 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Adherence, Treatment
MeSH Terms: conditions — Treatment Adherence and Compliance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Women with hormone-sensitive early breast cancer: Women older than 18 years of age who have suffered from hormonally dependent breast cancer stages 0-III (from "in situ" to locally advanced breast cancer) according to the American Joint Committee on Cancer (AJCC) classification and have been undergoing adjuvant endocrine therapy for more than 3 months.
  Interventions: Drug: Survey using a questionnaire.

INTERVENTIONS:
Drug: Survey using a questionnaire. — An observational study conducted in a cross-sectional manner using a questionnaire.

SUMMARY:
Breast cancer is the most common type of cancer and the leading cause of cancer death in women. Adjuvant endocrine therapy (AET) reduces the risk of disease recurrence and mortality in women with hormone-dependent breast cancer. This cross-sectional study aims to investigate adherence to AET and identify factors associated with adherence in the Republic of Croatia. The level of adherence, beliefs about medicines, and quality of life with AET will be investigated with validated instruments in the form of an anonymous survey. Given the available data on suboptimal adherence to AET in Europe and globally, it is clear that there is a need for investigating adherence in Croatia which hasn't been done so far. Each country, population, and health system has its own characteristics, and understanding the experience of using AET and identifying associated psychosocial factors could help in developing specific interventions supporting women and improving AET adherence.

ELIGIBILITY:
Inclusion Criteria:

* women older than 18 years of age
* clinical diagnosis of hormone receptor positive early breast cancer stages 0-III according to the American Joint Committee on Cancer (AJCC) classification
* prescribed with adjuvant endocrine therapy for more than 3 months

Exclusion Criteria:

* advanced metastatic breast cancer, stage IV according to the American Joint Committee on Cancer (AJCC) classification
* other life-threatening illnesses
* mental disorders
* behavioral disorders caused by the use of psychoactive substances
* behavioral syndromes related to physiological disorders and physical factors
* cognitive impairment
* organic and symptomatic mental disorder
* schizophrenia
* disorders similar to schizophrenia
* delusional disorders
* personality disorders
* behavior disorders
* mental retardation
* psychological development disorders
* unspecified mental disorders
* Incapable of autonomously reaching decisions

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study population comprises women aged 18 and older who have been diagnosed with hormone-dependent breast cancer at stages 0-III, as per the American Joint Committee on Cancer (AJCC) classification. These women have been receiving adjuvant endocrine therapy for a duration exceeding 3 months.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2024-09-20 (Estimated); Study Completion 2024-09-20 (Estimated)

PRIMARY OUTCOMES:
Patient adherence to adjuvant endocrine therapy assessment: Measurement of the level of adherence to adjuvant endocrine therapy | Day 1.
  The overall aim of the study is to determine the proportion of women adherent to oral adjuvant endocrine therapy (AEL) after the diagnosis of breast cancer in Croatia, as well as to investigate the association between AEL adherence, medication beliefs, quality of life, sociodemographic, and clinical factors.

SECONDARY OUTCOMES:
Beliefs About Medicines | Day 1.
  Investigate medication beliefs using the Medication Beliefs Questionnaire (BMQ).
Prevalence of Treatment-Emergent Adverse Events as assessed by FACT-ES | Day 1.
  Examine the quality of life using the Quality of Life Questionnaire with endocrine symptoms (FACT-ES).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zagreb Faculty of Pharmacy and Biochemistry, Zagreb, Croatia